CLINICAL TRIAL: NCT01903135
Title: Prevalence of Obesity Hypoventilation Syndrome in Subjects With Obesity Referred to Clinical (Medical Analysis) Laboratories for Regular Follow-up
Brief Title: Prevalence of Obesity Hypoventilation Syndrome
Acronym: BIO-OHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-AGIR-02; 2013-A00744-41 (Other: ANSM)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2015-03

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: Obesity Hypoventilation Syndrome; Prevalence; Bicarbonate
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- [HCO3-] >= 27 mmol/L (Group 1) (Other): All obese patients with plasmatic[HCO3-] >= 27 mmol/L will be addressed to a pneumologist. The pneumology investigations will establish(or not) the diagnosis of OHS
  Interventions: Procedure: Blood test analysis in the clinical labs; Procedure: Pneumologist consult to establish the diagnosis of OHS
- [HCO3-]< 27mmol/L+pneumologist (Group 2) (Other): Among obese patients with serum [HCO3-]< 27 mmol/L, 300 randomized patients will be addressed to a pneumologist. The pneumology investigations will refute(or not)the diagnosis of OHS.
  Interventions: Procedure: Blood test analysis in the clinical labs; Procedure: Pneumologist consult to establish the diagnosis of OHS
- [HCO3-]< 27 mmol/L (Group 3) (Other): Obese patients with a [HCO3-]<27 mmol/L randomized to group 3 will receive usual medical follow-up (end of study)
  Interventions: Procedure: Blood test analysis in the clinical labs

INTERVENTIONS:
Procedure: Blood test analysis in the clinical labs — for specific measurement of plasmatic bicarbonate
Procedure: Pneumologist consult to establish the diagnosis of OHS — complete respiratory check-up: Arterial blood gases analysis, spirometry, anthropometry, polygraphy or polysomnography.
  Medical history, previous treatments.
  Arms: [HCO3-] >= 27 mmol/L (Group 1); [HCO3-]< 27mmol/L+pneumologist (Group 2)

SUMMARY:
Rationale of the "BIO-OHS" study (Prevalence of Obesity Hypoventilation Syndrome):

The overall prevalence of Obesity Hypoventilation Syndrome (OHS) has never been directly assessed in the general population. Actually, this prevalence has been assessed in patients referred to sleep clinics with a potential diagnosis of sleep-disordered breathing or in patients already diagnosed with sleep apnea. The purpose of this study is to determine the prevalence of Obesity Hypoventilation syndrome in obese patients referred to clinical laboratories for regular follow-up medical analysis.

DETAILED DESCRIPTION:
No additional description

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ans more
* BMI over 30 kg/M2
* Stable state (respiratory, metabolic and cardio-vascular) for the last 2 months
* Addressed to a clinical labs for a blood check-up whatever the prescription

Exclusion Criteria:

* No social security
* Non cooperative patient, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Obesity Hypoventilation Syndrome (OHS) in obese subjects referred to clinical laboratories for regular blood test analysis. | From date of inclusion until the end of the study currently planned (up to 2 years)
  OHS prevalence, validated by arterial blood gases analysis, will be assessed by the percentage of patients with OHS among all patients included in the study

SECONDARY OUTCOMES:
Sensitivity and specificity of plasmatic [HCO3-] to detect OHS | From date of inclusion to the end of the study currently planned (2 years)
  A ROC curve will determine if the threshold of 27 mmol/L has the best diagnostic value.
  Decision trees will show if the diagnostic value of plasmatic [HCO3-]could be optimized by a combination with other clinical parameters.
Prevalence of metabolic and cardiovascular comorbidities in patients with OHS | From date of inclusion to the end of the study currently planned (2 years)
  Prevalence will be estimated by the percentage and the confidence interval. Prevalences of metabolic and cardiovascular comorbidities among patients with OHS and without OHS will be compared by a KHI-2 test or Fisher Exact depends on the theorical number.
To determine which medical specialties referred patients with OHS to clinical labs | From date of inclusion to the end of the study currently planned (2 years)
  estimated by percentage
Incidence of serious health events at 1 and 2-year follow-up | From time of OHS diagnostic to 1 and 2-year follow-up
  Cardiovascular, metabolic and respiratory events (measured by percentages in OHS group and non-OHS group) will be compared by logistic regressions.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, Pr, PhD, Principal Investigator — University Hospital, Grenoble
Locations (5):
- France (5):
  - Cabinet de Pneumologie Grenoble SUD, Échirolles
  - Laboratoire MEDIBIO Les Cedres, Échirolles
  - Hôpital Michallon, Laboratoire EFCR et Sommeil, Grenoble
  - Cabinet de Pneumologie Perpignan, Perpignan
  - Laboratoire d'analyses medicales de Thuir, Thuir

IPD SHARING:
Plan to Share IPD: Undecided